CLINICAL TRIAL: NCT00080444
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study, Conducted Under In-House Blinding Conditions, to Examine the Safety, Tolerability, and Efficacy of Aprepitant for the Prevention of Chemotherapy-Induced Nausea and Vomiting Associated With Emetogenic Chemotherapy in Adolescent Patients
Brief Title: Study of Aprepitant (MK-0869) for Chemotherapy-Induced Nausea and Vomiting (CINV) in Adolescent Participants (MK-0869-097)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 0869-097; Formerly-0304AHEC; MK-0869-097 (Other: Merck Protocol Number); 2004_099 (Other: Telerx Protocol Number)
Record Dates: First submitted 2004-03-31; First posted 2004-04-02 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Vomiting
MeSH Terms: conditions — Vomiting | interventions — Aprepitant; Ondansetron; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1: Aprepitant (Experimental): Day 1: aprepitant 125 mg orally (PO), ondansetron 0.15 mg/kg x 3 doses intravenously (IV), dexamethasone 8 mg PO. Day 2: aprepitant 80 mg PO, ondansetron 0.15 mg/kg x 3 doses IV, dexamethasone 4 mg PO. Day 3: aprepitant 80 mg PO, dexamethasone 4 mg PO. Day 4: dexamethasone 4 mg PO. For 1 cycle and up to 9 subsequent optional cycles.
  Interventions: Drug: aprepitant; Drug: ondansetron; Drug: dexamethasone; Drug: placebo to dexamethasone; Drug: rescue medication
- Part 1: Standard Therapy (Active Comparator): Day 1: placebo to aprepitant 125 mg PO, ondansetron 0.15 mg/kg x 3 doses IV, dexamethasone 16 mg PO. Day 2: placebo to aprepitant 80 mg PO, ondansetron 0.15 mg/kg x 3 doses IV, dexamethasone 8 mg PO. Day 3: placebo for aprepitant 80 mg PO, dexamethasone 8 mg PO. Day 4: dexamethasone 8 mg PO. For 1 cycle; participants may receive open-label aprepitant for up to 9 subsequent optional cycles.
  Interventions: Drug: ondansetron; Drug: dexamethasone; Drug: placebo to aprepitant; Drug: rescue medication
- Part 2: Aprepitant (Active Comparator): Day 1: aprepitant 125 mg PO, ondansetron 0.15 mg/kg x 3 doses IV, dexamethasone 8 mg PO. Day 2: aprepitant 80 mg PO, ondansetron 0.15 mg/kg x 3 doses IV, dexamethasone 4 mg PO. Day 3: aprepitant 80 mg PO, dexamethasone 4 mg PO. Day 4: dexamethasone 4 mg PO. For up to 10 cycles.
  Interventions: Drug: aprepitant; Drug: ondansetron; Drug: dexamethasone; Drug: placebo to dexamethasone; Drug: rescue medication

INTERVENTIONS:
Drug: aprepitant — aprepitant capsules
  Arms: Part 1: Aprepitant; Part 2: Aprepitant
Drug: ondansetron — ondansetron IV preparation
Drug: dexamethasone — dexamethasone tablets
Drug: placebo to aprepitant — Matching placebo to aprepitant capsules
  Arms: Part 1: Standard Therapy
Drug: placebo to dexamethasone — Matching placebo to dexamethasone tablets
  Arms: Part 1: Aprepitant; Part 2: Aprepitant
Drug: rescue medication — Participants are allowed to take rescue medication throughout for nausea or vomiting. At the discretion of the investigator, participants are provided with a prescription for rescue medications. Recommended rescue medications are: 5-HT3 antagonists, phenothiazines, butyrophenones, benzamides, corticosteroids, benzodiazepines, domperidone, H1-receptor antagonist, and piperazine derivatives.

SUMMARY:
This study is being conducted to demonstrate that aprepitant (MK-0869) prevents nausea and vomiting caused by emetogenic cancer chemotherapy in adolescent participants. Participants treated with emetogenic cancer chemotherapies that include either cisplatin, cyclophosphamide, or carboplatin, or participants who experienced nausea and/or vomiting when treated with a previously administered chemotherapy regimen that is planned to be repeated will be enrolled in this study. In the double-blind Part 1 of this study, enrolled participants will be randomized to receive either aprepitant or standard therapy. In Part 2 of this study, enrolled participants will receive open-label aprepitant.

DETAILED DESCRIPTION:
The duration of treatment is the first 4 days of one 28-day cycle (Cycle 1). Participants who successfully complete Cycle 1 may be eligible to participate for 9 subsequent optional, open-label, 28-day cycles.

ELIGIBILITY:
Inclusion Criteria:

* Cycle 1: Participant is to be treated with an emetogenic chemotherapy regimen that includes either cisplatin, cyclophosphamide, or carboplatin, for a documented malignancy. OR Participant did not tolerate a previously administered chemotherapy regimen, for a documented malignancy, secondary to nausea and/or vomiting that is planned to be repeated.
* Cycle 1: Participant has Karnofsky score ≥60
* Cycle 1: Participant has a predicted life expectancy of ≥3 months

Exclusion Criteria:

* Cycle 1: Participant will receive stem cell rescue therapy in conjunction with course of chemotherapy.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2004-04; Primary Completion 2006-09 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Experience Study-drug-related Adverse Events (Cycle 1) | Up to 14 days after last dose of anti-emetic therapy in Cycle 1 (Up to 18 days)

SECONDARY OUTCOMES:
Percentage of Participants Who Experience a Complete Response (CR) to Anti-emetic Therapy (Cycle 1) | Up to 120 hours after initiation of emetogenic chemotherapy in Cycle 1
Percentage of Participants Who Experience Absence of Nausea (Cycle 1) | Up to 120 hours after initiation of emetogenic chemotherapy in Cycle 1
Percentage of Participants Who Experience Absence of Vomiting (Cycle 1) | Up to 120 hours after initiation of emetogenic chemotherapy in Cycle 1
Percentage of Participants Who Experience Serious Adverse Events (Cycles 2-10) | Up to 14 days after last dose of anti-emetic therapy in Cycles 2-10 (Up to 10.5 months)
Percentage of Participants Who Experience Study-drug-related Adverse Events (Cycles 2-10) | Up to 14 days after last dose of anti-emetic therapy in Cycles 2-10 (Up to 10.5 months)
Percentage of Participants Who Discontinue Study Due to Study-drug-related Adverse Events (Cycles 2-10) | Up to Day 4 of Cycles 2-10 (Up to 10 months)
Percentage of Participants Who Experience Serious Adverse Events (Cycle 1) | Up to 14 days after last dose of anti-emetic therapy in Cycle 1 (Up to 18 days)
Percentage of Participants Who Experience Serious Study-drug-related Adverse Events (Cycle 1) | Up to 14 days after last dose of anti-emetic therapy in Cycle 1 (Up to 18 days)
Percentage of Participants Who Discontinue Study Due to Study-drug-related Adverse Events (Cycle 1) | Up to Day 4 of Cycle 1
Aprepitant Plasma Drug Concentration Profiles and Pharmacokinetics | Up to 24 hours after first dose of aprepitant

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Gore L, Chawla S, Petrilli A, Hemenway M, Schissel D, Chua V, Carides AD, Taylor A, Devandry S, Valentine J, Evans JK, Oxenius B; Adolescent Aprepitant in Cancer Study Group. Aprepitant in adolescent patients for prevention of chemotherapy-induced nausea and vomiting: a randomized, double-blind, placebo-controlled study of efficacy and tolerability. Pediatr Blood Cancer. 2009 Feb;52(2):242-7. doi: 10.1002/pbc.21811. PMID 18985740